CLINICAL TRIAL: NCT00496548
Title: Urinary PGE-M, A Metabolite of PGE2: A Novel Biomarker of Crohn's Disease Activity
Brief Title: Urinary Prostaglandin E Metabolite (PGE-M), A Metabolite of Prostaglandin E2 (PGE2): A Novel Biomarker of Crohn's Disease Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Principal Investigator, David Schwartz, Principal Investigator, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Urinary PGE-M CD
Record Dates: First submitted 2007-07-02; First posted 2007-07-04 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Fecal calprotectin and urinary PGE-M levels will be tested on all participants.
  Interventions: Procedure: Fecal calprotectin; Procedure: Urinary PGE-M Level

INTERVENTIONS:
Procedure: Fecal calprotectin — Fecal calprotectin levels obtained and compared to urinary PGE-M and serum C-reactive protein (CRP) levels.
Procedure: Urinary PGE-M Level — Urinary PGE-M level obtained and compared to fecal calprotectin and serum CRP levels.

SUMMARY:
The purpose of this study is to determine whether urinary PGE-M levels correlate with Crohn's disease activity and to compare how well urinary PGE-M correlates with other non-invasive biomarkers of disease activity such as C-reactive protein (CRP) and fecal calprotectin.

DETAILED DESCRIPTION:
The available clinical measures of Crohn's disease activity can be overly influenced by functional symptoms. Placebo response rates in clinical trials are high. Several non-invasive biomarkers are currently available for assessing inflammatory bowel disease (IBD) disease activity including erythrocyte sedimentation rate, C-reactive protein and fecal calprotectin. Although these markers hold some promise, their performance is less than ideal. What is needed is a simple, non-invasive, biologic measure of Crohn's disease.

Cyclooxygenase-2 (COX-2) is involved in prostaglandin E2 (PGE2) synthesis and is expressed in epithelial inflammatory conditions and some cancers. We have developed an assay to quantify the major urinary metabolite of PGE2, PGE-M. PGE-M has been previously shown to be elevated in the urine of patients with advanced colorectal neoplasia relative to controls.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient male or female 18 years or older
* Confirmed diagnosis of Crohn's disease
* Informed consent obtained
* Able to give blood, urine and stool samples
* Willing to undergo a diagnostic colonoscopy as part of routine Crohn's disease care

Exclusion Criteria:

* Unable to give consent
* Ulcerative colitis
* Does not meet inclusion criteria
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2007-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Urine for PGE-M levels | Day of colonoscopy procedure

SECONDARY OUTCOMES:
Blood for C-reactive protein (CRP) levels | Day 1
Stool for fecal calprotectin | Prior to colonoscopy procedure (before beginning bowel prep)
Routine colonoscopy for assessment of disease activity | 1-3 weeks from consent
Harvey-Bradshaw index disease activity score | Day of colonoscopy procedure

CONTACTS AND LOCATIONS:
Overall Officials: David A. Schwartz, MD, Principal Investigator — Vanderbilt University
Locations (1):
- GI Clinical Research; Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No